CLINICAL TRIAL: NCT04900194
Title: The Effect of Mindfulness-based Sexual Counseling on Sexual Distress, Attitudes Towards Sexuality and Body Image Concerns in Pregnant Women
Brief Title: The Effect of Mindfulness-based Sexual Counseling on Sexual Distress in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sıdıka Özlem CENGİZHAN, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-786
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Counseling
Keywords: pregnancy; mindfulness; sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSC group (Experimental): counseling group
  Interventions: Behavioral: mindfulness-based sexual counseling
- Control group (No Intervention): standard care group

INTERVENTIONS:
Behavioral: mindfulness-based sexual counseling — Mindfulness-based sexual counseling was planned as 2 sessions per week for 4 weeks, in total 8 sessions. Each session lasted 30-40 minutes on average. The sessions were carried out individually by determining the appropriate days of pregnant women in the pregnancy class.In the study, the meditation techniques of the Mindfulness Therapy constituted the backbone/framework of the psychoeducation program. Body and breath, body scanning, mindfulness movement and three-minute respiration techniques were practiced during the psychoeducation program, practically every session in accordance with the researchers' directives.
  Arms: MBSC group

SUMMARY:
The study was conducted in order to determine the effect of mindfulness-based sexual counseling on sexual distress, attitude towards sexuality and body image concerns in pregnant women. The research was planned in a randomized controlled experimental design.The sample consisted of the pregnant women who applied to the pregnant class at the time of the study and met the inclusion criteria. Female Sexual Distress Scale-Revised, Attitude towards Sexuality in Pregnancy Scale, Body Image Concerns During Pregnancy Scale were used. In the study, the pregnant women in the experimental group were given mindfulness-based sexual counseling by the researcher. Mindfulness-based sexual counseling was planned as 2 sessions per week for 4 weeks, in total 8 sessions. Each session lasted 30-40 minutes on average. First of all, Pregnancy Introduction Form, Attitude towards Sexuality in Pregnancy Scale, Female Sexual Distress Scale-Revised and Body Image Concerns in Pregnancy Scale were applied to the pregnant women in the experimental and control groups. The experimental group was given mindfulness-based sexual counseling for 4 weeks by the researcher. At the end of the mindfulness-based sexual counseling, the experimental group and the control group at the same time, were applied to the experimental group and the control group at the same time, the Female Sexual Distress Scale-Revised, Attitude towards Sexuality in Pregnancy Scale, and the Body Image Worries During Pregnancy Scale.

DETAILED DESCRIPTION:
The research was planned in a randomized controlled experimental design.The sample consisted of the pregnant women who applied to the pregnant class at the time of the study and met the inclusion criteria. In the power analysis used to determine the sample size, the 5% error level, the 95% confidence interval at the bilateral significance level, the 80% ability to represent the universe and the sexual distress mean score of 31.3 (standard deviation 10.9) in women. Assuming that 67 pregnant women were calculated for each group (67 experiments, 67 controls). Pregnancy Identification Form, Female Sexual Distress Scale-Revised, Attitude towards Sexuality in Pregnancy Scale, Body Image Concerns During Pregnancy Scale were used. In the study, the pregnant women in the experimental group were given mindfulness-based sexual counseling by the researcher. Mindfulness-based sexual counseling was planned as 2 sessions per week for 4 weeks, in total 8 sessions. Each session lasted 30-40 minutes on average. First of all, Pregnancy Introduction Form, Attitude towards Sexuality in Pregnancy Scale, Female Sexual Distress Scale-Revised and Body Image Concerns in Pregnancy Scale were applied to the pregnant women in the experimental and control groups. The experimental group was given mindfulness-based sexual counseling for 4 weeks by the researcher. At the end of the mindfulness-based sexual counseling, the experimental group and the control group at the same time, were applied to the experimental group and the control group at the same time, the Female Sexual Distress Scale-Revised, Attitude towards Sexuality in Pregnancy Scale, and the Body Image Worries During Pregnancy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Communicating,
* Over the age of 18,
* Pregnancy week between 10-28 weeks,
* Scoring 11.5 points and above according to the Female Sexual Distress Scale-Revised,

Exclusion Criteria:

* Sexual distress before pregnancy,
* Pregnant women with psychological diagnosis according to records.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Female Sexual Distress | Change from Female Sexual Distress at 4 weeks
  It is used to identify women with and without sexual dysfunction, evaluating subjective stress and psychological effects associated with sexual function. Responses to the items in the five-point Likert scale consist of never (0), rarely (1), sometimes (2), often (3), or always (4). The lowest score that can be obtained from the scale is 0, the highest score is 52. Higher scores indicate higher levels of sexual distress.

SECONDARY OUTCOMES:
The Scale of Attitude towards Sexuality in Pregnancy | Change from Attitude towards Sexuality at 4 weeks
  The items contain cognitive, affective and behavioral components of sexual attitude. The scale has three sub-dimensions; "Anxiety Towards Sexual Intercourse During Pregnancy", "Beliefs and Values Towards Sexuality During Pregnancy", "Confirming Sexuality During Pregnancy". The total score that can be obtained from the total score of the scale is the lowest 34 and the highest 170. The increase in the total score obtained from ATSPS indicates that the attitudes towards sexuality during pregnancy are positive, and the decrease in the total score indicates that the attitudes towards sexuality during pregnancy are negative.
Body Image Worries in Pregnancy Scale | Change from Body Image Worries at 4 weeks
  The scale consists of 4 sub-dimensions. Sub-dimensions of the scale Avoidance, Social worries, Worries about weight gain, Future worries, physical appearance concerns.The highest score to be obtained from the scale is 115, the lowest score is 23.An increase in the total score of the scale indicates that concerns about body image are high during pregnancy, while a decrease indicates that concerns about body image during pregnancy are low.

CONTACTS AND LOCATIONS:
Overall Officials: Sıdıka Özlem Cengizhan, Msc, Principal Investigator — Inonu University
Locations (1):
- Faculty of Health Science, Malatya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data were not shared

REFERENCES:
- [Result] Nezamnia M, Iravani M, Bargard MS, Latify M. Effectiveness of cognitive-behavioral therapy on sexual function and sexual self-efficacy in pregnant women: An RCT. Int J Reprod Biomed. 2020 Aug 19;18(8):625-636. doi: 10.18502/ijrm.v13i8.7504. eCollection 2020 Aug. PMID 32923929
- [Result] Brotto LA, Basson R, Luria M. A mindfulness-based group psychoeducational intervention targeting sexual arousal disorder in women. J Sex Med. 2008 Jul;5(7):1646-59. doi: 10.1111/j.1743-6109.2008.00850.x. PMID 18507718
- [Derived] Cengizhan SO, Ucar T. The Effect of Mindfulness-Based Sexual Counseling on Sexual Distress, Attitude Toward Sexuality, and Body Image Concerns in Pregnant Women: A Randomized Controlled Trial. J Midwifery Womens Health. 2023 Sep-Oct;68(5):611-618. doi: 10.1111/jmwh.13518. Epub 2023 Jun 9. PMID 37294101